CLINICAL TRIAL: NCT06558695
Title: Comparison of TIVA and Sevoflurane: Affirming Hemodynamic, Respiratory, and Neuromonitoring Stability in Prone Position Spinal Surgeries
Brief Title: Stability Comparison of TIVA and Sevoflurane in Prone Spinal Surgery(TIVA:Total Intravenous Anesthesia)
Acronym: TIVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, YÜCEL YÜCE, Associate Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: SaglikBilimleriU-KLKSH-Anes-01
Record Dates: First submitted 2024-08-12; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Spinal Stenosis, Lumbosacral Region
Keywords: Total intravenous anesthesia; Sevoflurane; Respiratory mechanics,; Hemodynamic parameters; Spinal surgery; Prone position
MeSH Terms: conditions — Spinal Stenosis | interventions — Sevoflurane

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial involved 52 patients scheduled for lumbar spine surgery under general anesthesia. Participants were randomly allocated to either the TIVA group (n=26) or the sevoflurane group (n=26). Measurements of respiratory mechanics, including peak airway pressure (Ppeak), mean airway pressure (Pmean), positive end-expiratory pressure (PEEP), end-tidal CO2 (ETCO2), tidal volume (VT), respiratory rate (RR), and minute ventilation (MV), were taken at various intervals. Hemodynamic parameters such as systolic and diastolic blood pressures and heart rate were continuously monitored.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were randomly assigned to one of two groups using a computer-generated list: the Sevoflurane group (Sevo group) and the Total Intravenous Anesthesia group (TIVA group), each comprising 26 patients. The assignment and subsequent anesthesia management were conducted in a double-blinded manner, ensuring that neither the patients nor the clinicians administering the treatments or assessing the outcomes were aware of the group allocations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevoflurane Group (Active Comparator): In the Sevoflurane group, general anesthesia was maintained with sevoflurane at 0.8-1.0 minimum alveolar concentration (MAC).
  Interventions: Drug: Sevoflurane
- TIVA group (Active Comparator): In the TIVA (Total Intra Venous Anesthesia) group, a combination of propofol (50-150 μg/kg/min) and remifentanil (0.02-0.2 μg/kg/min) was used for general anesthesia instead of inhalational agents.
  Interventions: Drug: TIVA

INTERVENTIONS:
Drug: Sevoflurane — Sevoflurane was managed for maintenance of the general anestesia during spinal surgeries
  Arms: Sevoflurane Group
Drug: TIVA — TIVA was managed for maintenance of the general anesthesia during spinal surgeries
  Other Names: Total Intra Venous Anesthesia
  Arms: TIVA group

SUMMARY:
Key Points:

1. Objective:

   o To compare the effects of Total Intravenous Anesthesia (TIVA) and sevoflurane anesthesia on respiratory mechanics, hemodynamic parameters, and neuromonitoring during prone position spinal surgeries.
2. Methodology:

   * A randomized controlled trial involving 52 patients scheduled for lumbar spine surgery, randomly assigned to either TIVA or sevoflurane groups.
   * Respiratory and hemodynamic parameters were measured at various time points.
3. Results:

   * No significant differences were found between the TIVA and sevoflurane groups in terms of respiratory mechanics or hemodynamic stability.
   * Both anesthesia techniques maintained stable intraoperative conditions.
4. Clinical Implications:

   * Anesthesiologists can flexibly choose between TIVA and sevoflurane based on patient-specific factors and surgical requirements.
   * TIVA may be preferred in surgeries with high neurological risk due to its compatibility with neuromonitoring.
5. Future Research:

   * Studies with broader patient populations and long-term outcomes are needed to further refine anesthesia management strategies.
   * Research on the environmental impact and cost-effectiveness of anesthesia techniques is also important.

DETAILED DESCRIPTION:
This study aims to evaluate the impact of total intravenous anesthesia (TIVA) versus sevoflurane anesthesia on respiratory mechanics and hemodynamic parameters during spinal surgery performed in the prone position. Anesthesia management for spinal surgeries in the prone position is particularly challenging due to significant physiological changes. Identifying the effects of different anesthesia techniques is essential to enhance patient outcomes and ensure intraoperative stability. This randomized controlled trial involved 52 patients scheduled for lumbar spine surgery under general anesthesia. Participants were randomly allocated to either the TIVA group (n=26) or the sevoflurane group (n=26). Measurements of respiratory mechanics, including peak airway pressure (Ppeak), mean airway pressure (Pmean), positive end-expiratory pressure (PEEP), end-tidal CO2 (ETCO2), tidal volume (VT), respiratory rate (RR), and minute ventilation (MV), were taken at various intervals. Hemodynamic parameters such as systolic and diastolic blood pressures and heart rate were continuously monitored.

ELIGIBILITY:
Inclusion Criteria:

* The study included male and female patients aged 18 to 65 years who were scheduled for lumbar spine surgery under general anesthesia. Patients were categorized based on the American Society of Anesthesiologists (ASA) physical status levels I, II, and III.

Exclusion Criteria:

* Diagnosis of asthma or chronic obstructive pulmonary disease (COPD)
* Major cardiac conditions, such as recent myocardial infarction or a left ventricular ejection fraction (EF) less than 55%
* Atrioventricular blocks of second and third degrees
* Allergies to any drugs
* Severe neurological disorders
* History of sedative or opioid use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
PEEP | 5, 15, and 30 minutes after positioning in the prone position
  positive end-expiratory pressure
ETCO2 | 5, 15, and 30 minutes after positioning in the prone position
  end-tidal carbon dioxide
VT | 5, 15, and 30 minutes after positioning in the prone position
  tidal volume
Ppeak | 5, 15, and 30 minutes after positioning in the prone position
  peak airway pressure
Pmean | 5, 15, and 30 minutes after positioning in the prone position
  mean airway pressure
RR | 5, 15, and 30 minutes after positioning in the prone position
  Respiratory Rate
MV | 5, 15, and 30 minutes after positioning in the prone position
  Minute volume
Cdyn | in the supine position after intubation and in the prone position at the 30th minute
  Dynamic. compliance
PaO2/FiO2 | in the prone position at the 30th minute
  Partial Oxygen pressure/traction of inspired oxygen
Vd/Vt | in the prone position at the 30th minute
  dead space/tidal volume

SECONDARY OUTCOMES:
HR | 5, 15, and 30 minutes after positioning in the prone position
  Heart Rate
SBP | 5, 15, and 30 minutes after positioning in the prone position
  Systolic Blood Pressure
DBP | 5, 15, and 30 minutes after positioning in the prone position
  Diastolic BloodPressure

CONTACTS AND LOCATIONS:
Overall Officials: Yücel Yüce, MD,Assoc Prf, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Saglik Bilimleri Universitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No